CLINICAL TRIAL: NCT06163209
Title: High-resolution Point of Care Ultrasonography in the Diagnosis of Nasal Fractures: a 10-step Protocol
Brief Title: Ultrasonography in the Diagnosis of Nasal Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Grzegorz Śmigielski, Principal Investigator, Medical University of Gdansk
Other Study IDs: NFUS2023
Record Dates: First submitted 2023-11-29; First posted 2023-12-08 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Nasal Bone Fracture; Nasal Injury; Facial Injuries; Nasal Deformity, Acquired; Nose; Wound
Keywords: high-resolution ultrasonography; point-of-care ultrasonography; nasal fracture
MeSH Terms: conditions — Facial Injuries; Nose Deformities, Acquired; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Suspected nasal fracture: Patients with a history of recent nasal trauma.
  Interventions: Diagnostic Test: Nasal Ultrasonography; Diagnostic Test: Computed Tomography Scan of the Face

INTERVENTIONS:
Diagnostic Test: Nasal Ultrasonography — Ultrasonography of the external nose will be performed with the use of a high-resolution transducer (Clarius L20HD3 8-20 MHz) and a 3mm-thick disposable gel pad, according to the following protocol:
  1. Sagittal plane, along the most prominent part of nasal dorsum.
  2. Transverse plane, level of nasion.
  3. Transverse plane, level of intercanthal line.
  4. Transverse plane, level of rhinion.
  5. Along inferior border of the right nasal bone.
  6. Along inferior border of the left nasal bone.
  7. Along medial part of the right orbital rim below frontomaxillary suture.
  8. Along medial part of the right orbital rim below frontomaxillary suture.
  9. Along the line connecting right frontomaxillary suture and the tip of the nose.
  10. Along the line connecting left frontomaxillary suture and the tip of the nose.
  At each location the transducer position will be adjusted until it is held perpendicular to the bone surface and a single image will be saved for further assessment.
  Other Names: High resolution 10-point ultrasonography of the external nose.
Diagnostic Test: Computed Tomography Scan of the Face — A standard computed tomography scan of the face will be performed and the following areas will be assessed by an experienced radiologist:
  1. Bony part of the nasal septum
  2. Left nasal bone - part proximal to the intercanthal line
  3. Right nasal bone - part proximal to the intercanthal line
  4. Left nasal bone - part distal to the intercanthal line
  5. Right nasal bone - part distal to the intercanthal line
  6. Frontal process of the left maxilla
  7. Frontal process of the right maxilla
  Other Names: A computed tomography covering the whole facial skeleton and a skull base.

SUMMARY:
The purpose of this cross-sectional prospective observational study is to determine the efficacy of high-resolution ultrasonography in identifying and characterizing nasal bone fractures in adult patients with recent facial trauma. The primary questions it aims to answer are:

* Can high-resolution ultrasonography effectively detect nasal bone fractures?
* Is high-resolution ultrasonography capable of indirectly detecting septal fractures?
* What are the specificity and sensitivity of high-resolution ultrasonography in comparison to computed tomography scan?

Participants will undergo examination and treatment in accordance with current standards for nasal fracture management. Additionally, high-resolution ultrasonography will be performed during the initial physical examination, preceding any therapeutic interventions.

DETAILED DESCRIPTION:
BACKGROUND

The bony and cartilaginous skeleton of the external nose is exceptionally prone to injury, due to its fragile structure and protruding, tent-like shape. As the cartilages are able to bend under pressure, the impact of trauma is usually transferred to the thinnest, distal parts of nasal bones, where they overlap the lateral cartilages forming a junction called the keystone region. This location plays a major role in supporting the cartilaginous skeleton and, at the same time, is most likely to be fractured. Similarly, the cartilaginous nasal septum is able to bend, which is the reason why trauma to the distal nasal bones frequently continues along anterior borders of the perpendicular plate of the ethmoid and vomer, creating a complex, C-shaped septal fracture. These pathomechanisms of nasal fracture explain its possible significant negative influence on the function and aesthetics of the nose. Early nasal fracture detection and treatment is critical for avoiding complications. Clinical examination is considered a gold standard for the diagnosis. Imaging tests are of secondary importance, as their clinical application in this condition has many disadvantages. A commonly applied plain radiograph of the nose was proven not to be cost efficient due to high percentage of false results. A computed tomography scan (CT) has a satisfactory sensitivity and specificity, but is relatively expensive, causes radiation exposure and provides images of limited resolution, which may fail to reveal subtle fracture lines.

Several studies have shown high-resolution ultrasonography (HRUS) to be a safe and efficient method for nasal fracture diagnosis. However, the use of this modality in a clinical setup has not become common, despite over 20-year history of publications supporting its efficacy. Potential factors contributing to this circumstance include a lack of a standardized examination protocol, a difficult ultrasonography image acquisition and a clinician's reluctance to use a full-sized device in an otolaryngology medical office.

The aim of this study is to assess the efficacy of a standardized 10-step point-of-care ultrasonography in the diagnosis of nasal fractures.

STUDY DESIGN

This cross-sectional prospective study will be conducted between December 1, 2023, and December 1, 2024, at the University Clinical Centre in Gdańsk, in accordance with the Helsinki Declaration and with approval from the institutional bioethics committee for scientific research (No: KB/625/2023).

Patients who have presented to the emergency department with nasal trauma sustained within the 14 days preceding their consultation will be enrolled in the study. Exclusion criteria will include extensive facial trauma, a history of nasal fracture, surgical interventions (e.g. rhinoplasty, frontal/ethmoid sinus surgery), or minor invasive procedures (e.g. hyaluronic acid filler, thread lifting) in the examined area.

A CT scan of the face and HRUS protocol will be performed before any interventions are undertaken.

A total of 50 patients is anticipated.

The collected data will include medical history, physical examination, CT scan of the face and HRUS of the nose.

Ultrasonography of the external nose will be performed with the use of a high-resolution transducer (Clarius L20HD3 8-20 MHz) and a 3mm-thick disposable gel pad, according to the 10-step protocol. At each location, the transducer position will be adjusted with rocking and tilting movements until it is held perpendicular to the bone surface, which provides optimal image quality, and a single image will be saved for further assessment. Images obtained at each location will be assessed for five different findings.

A standard computed tomography scan of the face will be performed. Each of 7 specific areas will be assessed by an experienced radiologist for a diclocated or non-dislocated nasal fracture.

DATA ANALYSIS

Statistical analysis of the data will be performed using the R language. A variable marked as a "final diagnosis established by the consulting clinician" will be considered a reference point for calculating the sensitivity and specificity of methods. For this purpose, a McNeymar chi-square test and Cohen's Kappa will be used.

Records lacking the final diagnosis or any part of the HRUS protocol will be excluded from the study.

The database will be anonymised.

The source data and the database verification will be performed collectively by the authors following the addition of every 10 new records.

ELIGIBILITY:
Inclusion Criteria:

* nasal trauma during the 14 days preceding examination

Exclusion Criteria:

* extensive facial injuries
* history of surgical or non-surgical interventions in the examined area
* history of nasal fracture
* refusal to participate, inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a history of recent facial trauma involving external nose. Patients with no history of surgical or non-surgical interventions in the examined area eg. rhinoplasty, hyaluronic acid filler, external approach frontal/ethmoid sinus surgery as well as no history of nasal fracture.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Nasal Ultrasonography: a 10-step protocol. | Each participant will be assessed once, within 14 days of the nasal trauma.
  Images obtained at each location will be assessed for the following five findings:
  1. isolated bone discontinuity
  2. misalignment of the bone surface without displaced fracture edges
  3. misalignment of the bone surface with displaced fracture edges
  4. dislocated minor bone fragment (largest dimension under 2 mm)
  5. soft tissue haematoma
  There will be 50 variables in total, marked as a combination of location (number 1-10) and finding (a-e) e.g. 1a, 1b, 1c, 1d, 1e, 2a, 2b, 2c ,2d.
  Variables will be dichotomous, with possible values of P (positive), N (negative) and N/A (not to be assessed).

SECONDARY OUTCOMES:
Computed Tomography of the Face | Each participant will be assessed once, within 14 days of the nasal trauma.
  Each of 7 anatomical areas will be assessed for one of two findings:
  1. non-displaced fracture
  2. displaced fracture
  There will be 14 variables in total, marked as a combination of location (number 1-7) and finding (a-b) e.g. 1a, 1b, 2a, 2b, 3a, 3b.
  Variables will be dichotomous, with possible values of P (positive), N (negative) and N/A (not to be assessed).
Clinical features | Each participant will be assessed once, within 14 days of the nasal trauma.
  Following clinical data associated with present nasal trauma will be collected and entered into the database as variables:
  * time period since the injury
  * epistaxis
  * nasal obstruction
  * crepitus or palpable mobility of bone fragments
  * swelling of the nasal pyramid
  * nasal pyramid asymmetry - absent before trauma
  * septal deviation - absent before trauma
  * fracture reposition attempt
  * improvement after reposition
  Variables will be dichotomous, with possible values of P (positive), N (negative) and N/A (not to be assessed), except for time period, which will be a number in the range from 0 to 14.

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Śmigielski, M.D., Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdańsk, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan will be shared upon request, including individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
  Proposals should be directed to "g.smigielski@gumed.edu.pl". To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 36 months following article publication.
Access Criteria: For individual participant data meta-analysis. Proposed use of the data should have been approved by an independent review committee.

REFERENCES:
- [Background] Gokcen E, Savrun A, Kusdogan M, Caltekin I, Albayrak L, Atik D, Vural S, Savrun ST, Yildirim G. Ability of Bedside Ultrasonography to Detect Pediatric Nasal Bone Fractures. Laryngoscope. 2021 Jun;131(6):1398-1403. doi: 10.1002/lary.29168. Epub 2020 Oct 3. PMID 33009831
- [Background] Astaraki P, Baghchi B, Ahadi M. Diagnosis of acute nasal fractures using ultrasound and CT scan. Ann Med Surg (Lond). 2022 May 26;78:103860. doi: 10.1016/j.amsu.2022.103860. eCollection 2022 Jun. PMID 35734733
- [Background] Shigemura Y, Ueda K, Akamatsu J, Sugita N, Nuri T, Otsuki Y. Ultrasonographic Images of Nasal Bone Fractures with Water Used as the Coupling Medium. Plast Reconstr Surg Glob Open. 2017 May 30;5(5):e1350. doi: 10.1097/GOX.0000000000001350. eCollection 2017 May. PMID 28607870
- [Background] Westfall E, Nelson B, Vernon D, Saltagi MZ, Mantravadi AV, Schmalbach C, Ting JY, Shipchandler TZ. Nasal bone fractures and the use of radiographic imaging: An otolaryngologist perspective. Am J Otolaryngol. 2019 Nov-Dec;40(6):102295. doi: 10.1016/j.amjoto.2019.102295. Epub 2019 Sep 9. PMID 31526629
- [Background] Hwang K, Jung JS, Kim H. Diagnostic Performance of Plain Film, Ultrasonography, and Computed Tomography in Nasal Bone Fractures: A Systematic Review. Plast Surg (Oakv). 2018 Nov;26(4):286-292. doi: 10.1177/2292550317749535. Epub 2018 Jan 9. PMID 30450348
- [Background] Caglar B, Serin S, Akay S, Yilmaz G, Torun A, Adibelli ZH, Parlak I. The accuracy of bedside USG in the diagnosis of nasal fractures. Am J Emerg Med. 2017 Nov;35(11):1653-1656. doi: 10.1016/j.ajem.2017.05.015. Epub 2017 May 18. PMID 28552270
- [Background] Lee IS, Lee JH, Woo CK, Kim HJ, Sol YL, Song JW, Cho KS. Ultrasonography in the diagnosis of nasal bone fractures: a comparison with conventional radiography and computed tomography. Eur Arch Otorhinolaryngol. 2016 Feb;273(2):413-8. doi: 10.1007/s00405-015-3595-8. Epub 2015 Mar 8. PMID 25749616
- [Background] Hoffmann JF. An Algorithm for the Initial Management of Nasal Trauma. Facial Plast Surg. 2015 Jun;31(3):183-93. doi: 10.1055/s-0035-1555618. Epub 2015 Jun 30. PMID 26126215
- [Background] Gossner J. Sonography of the nasal cartilage: technique and normal anatomy. J Ultrasound. 2014 Aug 5;17(4):317-9. doi: 10.1007/s40477-014-0123-4. eCollection 2014 Dec. PMID 25368692
- [Background] Jecker P. [Diagnostic use of ultrasound for examination of the nose and the paranasal sinuses]. Ultraschall Med. 2005 Dec;26(6):501-6. doi: 10.1055/s-2005-857898. German. PMID 16453210